

**Official Title:** Assessing Cultures of Recovery in Tribal Communities – Research Core – Training Evaluation

**Brief Title:** First Face Training Evaluation in Tribal Communities

**Document:** First Face Evaluation Study Assent Form Age 14-17

**Date:** July 21<sup>st</sup>, 2023



# ASSENT FOR RESEARCH (14-17 year olds)

We try to make this form easy to understand. But it may have words or ideas that are not clear to you. Please ask a member of the study team to explain anything you do not understand. You may take this form home with you to discuss with family or friends before you decide whether to be in this research study.

| Study Title: First Face Training Evaluation Study | |
|---|---|
| Your name (Participant): | Today's Date: |
| Name of Investigators: Martina Whelshula, Ph.D., Debi A. LaPlante, Ph.D., Sarah E. Nelson, Ph.D., and Eric Louderback, Ph.D. | |

# Why am I here?

We want to talk to you and your parent(s)/guardian(s) about a research study being conducted by researchers from the Healing Lodge of the Seven Nations and Cambridge Health Alliance. The study is called the *First Face* Training Evaluation Study. Research is a special way to learn about something new. We would like you to take part because you live in one of the seven Tribal communities that work with the Healing Lodge. Taking part in this study is voluntary. You have the choice to take part or not. You may leave the study at any time for any reason.

#### Why is this study being done

This study is being done to evaluate a culturally grounded training program, xa?tus (meaning *First Face*) for Mental Health. This program will train you and other community members in how to recognize and respond to youth and adults experiencing mental health crises and ways to help them. We will have two training groups -- people who take *First Face* training this summer, and people who take the *First Face* training 6 months later. People in both groups will complete surveys before and after training about their knowledge and attitudes about mental health. The study will help us understand how well the *First Face* training program works and how to improve it.

## How many other people will take part in this study?

We hope to have at least 700 participants across seven Tribal Nations in Washington, Oregon, and Idaho – take part in this study. We are asking both teenagers and adults to participate.

## How long will I be in the study?

If you choose to participate, you will be in this study for up to 24 months. You will attend the *First Face* training, which will take about 8 hours, either this summer or 6 months later. You will also complete five surveys – one each at the beginning and end of the training, and three more online at six-month and 12-month intervals. Each survey will take 15-30 minutes to complete. You can stop being in the study at any time for any reason. But if you decide to stop, we encourage you to talk to one of us first.

## What do I have to do if I am in the study?

If you are in the study, you will:

- Participate in the First Face training, either this summer, or six months later.
- Complete five surveys, each of which is 15-30 minutes long. You will complete two of these surveys at the training. You will complete the other surveys online every 6 to 12 months. The surveys will ask you questions about your knowledge about mental health topics, your attitudes and beliefs about mental health, and how you feel about responding to mental health situations.

## What are the risks of taking part in the study?

If you take part in the study, you will participate in the *First Face* training and complete surveys. We do not anticipate any major risks from either of those activities. The following are possible minor risks:

- You might feel stressed or anxious during the training.
- The survey questions might make you feel embarrassed or stressed. You don't have to answer any questions you don't want to.
- Someone might tell other people what you say in the training or someone might see how you answered
  your surveys. We do everything we can to keep your information and your survey answers private and
  confidential.

#### What are the benefits of taking part in this study

You might not benefit directly from this training or study, but we hope the *First Face* training will be valuable to and give you knowledge and skills to help people in your community. What we learn from this study might help others in your community and beyond in the future.

# Will I get paid to be in this study?

You will be paid for your participation in the study. If you attend the *First Face* training and complete all five surveys, you will receive \$180 in gift cards. After each survey you complete, you will receive a gift card for \$20, \$30, \$40, or \$60, depending on the survey. You will only be paid for each survey that you complete.

## Do my parents/guardian need to know about this study?

Yes. We have told your parent(s)/guardian about this study. They know that we have invited you to take part. They will have to sign a permission form to allow you to be in this study.

## Who else will know I am in this study?

We will do our best to keep your information private. We will follow these guides:

- We will keep your surveys and data in a secure location.
- We will not include any information that could identify you (like your name) in any publication or report.
- We will remove all of your personal information from our study records 10 years after the study has been completed.

We will make every effort to keep your information private, but we cannot guarantee it. The Portland Area Institutional Review Board (IRB) is responsible for protecting the safety and welfare of people who take part in research studies in this region. IRB staff may ask to look at any research records to make sure the study team is following the laws and rules to protect you. Certain government agencies, including the Office for Human Research Protections, may also look at records that identify you.

Sometimes, we are required to share your study records with others, too, including:

- Other researchers conducting this study;
- The Portland Area Institutional Review Board (IRB). They are the group that makes sure that people who
  participate in research are kept safe;
- The government agency that gave us money to do the study.

#### **Costs**

If you take part in this study, there will be no cost to you.

## What if I am injured in this study?

It is very unlikely that you will be injured by participating in this study. If you do get hurt while in the study, no costs will be covered.

## What are my rights when I am in the study?

Being in this study is voluntary. You do not have to be in the study if you do not want to. You can stop being in the study at any time for any reason. But you should have your parent/guardian contact us if you decide to stop. If you decide not to take part or you decide to leave the study, you will not be punished.

# Who do I call if I have questions or problems?

If you have questions about this study, you can email a member of the study team. You can reach us Monday to Friday during regular business hours: Email: info@firstface.org You can also call the study team if you have an urgent question or concern: **Hannah Tomeo (Research Coordinator)** 509-795-8344 If you have questions about your rights as a study participant, you can call the Portland Area IRB Chair: IRB Chair - Thomas Weiser: 877-664-0604 Once you have made your decision, please check one of the boxes below and sign your name: Yes, I will take part in this research study No, I do not want to take part in this research study Signature of Adolescent Date Printed Name of Adolescent

Date

Printed Name of Researcher Obtaining Consent

Signature of Researcher Obtaining Consent